CLINICAL TRIAL: NCT04586621
Title: Evaluation of the Performance and Safety of the Atoldys/ Lexilens Glasses Developed to Improve the Reading of Dyslexic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ABEYE (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Atoldys/ Lexilens
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atoldys/ Lexilens - SHAM (Experimental)
  Interventions: Device: Atoldys/ Lexilens - SHAM
- SHAM- Atoldys/ Lexilens (Experimental)
  Interventions: Device: SHAM- Atoldys/ Lexilens

INTERVENTIONS:
Device: Atoldys/ Lexilens - SHAM — Atoldys/ Lexilens: glasses with specific light frequency SHAM: glasses with no frequency
  Arms: Atoldys/ Lexilens - SHAM
Device: SHAM- Atoldys/ Lexilens — SHAM: glasses with no frequency Atoldys/ Lexilens: glasses with specific light frequency
  Arms: SHAM- Atoldys/ Lexilens

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of a new medical device (Atoldys/ Lexilens glasses) on the improvement of reading skills of young dyslexic subjects.

DETAILED DESCRIPTION:
Dyslexia is defined as a specific learning disability that is characterized by reading difficulties, in the absence of intellectual disability, neurological or psychiatric disorder, uncorrected sensory disturbance (sight, hearing) or an educational deficiency.

Dyslexia appears in the child from the earliest stages of learning in the form of a difficulty in mastering the learning of reading. This disorder is manifested by a generally hesitant reading, slowed down, full of errors, requiring a lot of effort for the child and may impact his reading comprehension. The dyslexia-related deficiency is of variable intensity depending on the individual; it may be accompanied by calculus disorders (dyscalculia), oral language (dysphasia), motor coordination (dyspraxia) or attention disorders with or without hyperactivity. In nearly 40% of cases, a child affected by Dys disorders presents several learning disorders.

To date, the causes of dyslexia are not yet clearly established. The wide variety of symptoms and disorders associated with dyslexia does not facilitate the identification of precise neurobiological / psycho cognitive mechanisms. There are therefore several theories: phonological, visual, temporal, cerebellar or proprioceptive auditory processing.

Recently, following work published in 2017, an anatomical cause based on Maxwell's spots could also be a cause of dyslexia.

The aim of this study is to evaluate a new medical device (class I CE marked) to compensate this probable anatomical cause: the Atoldys/ Lexilens glasses

ELIGIBILITY:
Inclusion Criteria:

* Schooled in CM1, CM2 or 6ème,
* French mother tongue,
* For whom developmental dyslexia has been diagnosed by a health professional who specializes in this learning disorder,
* With near vision, without optical correction, equivalent to P5 or better according to the Parinaud scale (distance: 30-40 cm),
* Presenting an IQ ≥ 80 and ≤130 according to the WISC-V test performed by a psychologist,
* For whom a written consent was obtained regarding his study participation.

Exclusion Criteria:

* With medical history or presenting a neurological pathology,
* Presenting a developmental disorder (autism, ADHD, ...),
* Presenting hearing disorders,
* Presenting an astigmatism of more than one uncorrected diopter,
* Presenting other visual disorders,
* Any other condition that, in the opinion of health professionals, could impair its ability to complete the study or could pose a significant risk.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Reading performance aloud of a text with french E.L.FE Test | 1 day
  E.L.FE Test (=Evaluation de la Lecture en FluencE) - "Monsieur Petit" and "Le Géant égoïste" texts : percentile

SECONDARY OUTCOMES:
Reading performance aloud of isolated words with french BALE Test | 1 day
  BALE test (=Batterie Analytique de Langage Ecrit): percentile
Security: incidence of Adverse Events | 1 day
  By questioning the child & the speech therapist - evaluation of adverse effects due to glasses (Yes/ No): headache, nausea, dizziness, fatigue and eye fatigue. According to patient questioning and clinical exam, the Adverse Event Table will be completed (description, dates, severity, imputability, action,...).
Security: device deficiencies | 1 day
  By questioning the speech therapist - evaluation of deficiencies due to glasses: the device deficienciesTable will be completed (description, relation with adverse effect, taken measures,...).
Child's satisfaction regarding reading fluency and comprehension | 1 day
  Child interview with numeric scale (0-10) and yes/ no answer
Speech therapist's satisfaction regarding Securirty, Performance and Usability of glasses | 1 day
  speech therapist interview with 4 points - Likert scale (Very good, Good, Moderate, Bad)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Dr Laurence Derieux, Caen
  - Dr Luc-Marie Virlet, Faumont
  - CHU Rennes, Rennes